CLINICAL TRIAL: NCT05517486
Title: Parallel Study to Evaluate the Pharmacokinetics, Dose Proportionality, Safety and Tolerability of GTX-101 (Bupivacaine Hydrochloride Metered Dose Spray) and Subcutaneous Injectable Bupivacaine in Healthy Subjects
Brief Title: Single-dose to Evaluate the Pharmacokinetics of GTX-101 and Subcutaneous Injectable Bupivacaine in Healthy Subjects
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Grace Therapeutics Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: GTX-101-004
Record Dates: First submitted 2022-07-14; First posted 2022-08-26 (Actual); Last update posted 2023-01-23 (Actual); Status verified 2022-06

CONDITIONS: Postherpetic Neuralgia
MeSH Terms: conditions — Neuralgia, Postherpetic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- 50 mg GTX-101 (Experimental)
  Interventions: Drug: GTX-101
- 100 mg GTX-101 (Experimental)
  Interventions: Drug: GTX-101
- 200 mg GTX-101 (Experimental)
  Interventions: Drug: GTX-101
- Bupivacaine subcutaneous injection (Active Comparator)
  Interventions: Drug: Bupivacaine HCl subcutaneous injection

INTERVENTIONS:
Drug: GTX-101 — Bupivacaine HCl metered spray
  Other Names: Bupivacaine HCl metered spray
  Arms: 100 mg GTX-101; 200 mg GTX-101; 50 mg GTX-101
Drug: Bupivacaine HCl subcutaneous injection — Bupivacaine HCl, 50 mg/10 mL
  Arms: Bupivacaine subcutaneous injection

SUMMARY:
This is a single-center, randomized, single-dose, active-controlled study in healthy male and female subjects.

The study will enroll subjects to evaluate the PK of 3 dose strengths (50 mg, 100 mg and 200 mg) of GTX-101 compared to Subcutaneous injection in healthy adult subjects.

Blood samples for PK assessments will be collect at specified time points. Safety assessments will also be performed throughout the study.

ELIGIBILITY:
Inclusion Criteria:

* Provision of signed and dated informed consent form (ICF)
* Healthy adult male or female, aged 18 to 55 years, inclusive, at Screening
* Body mass index (BMI) within 18.0 kg/m2 to 30.0 kg/m2, inclusively at Screening
* Have no clinically significant diseases captured in the medical/surgical history or evidence of clinically significant findings on the physical examination (including vital signs), weight and/or clinical laboratory tests and/or ECG, as determined by an Investigator

Exclusion Criteria:

* History of significant hypersensitivity to bupivacaine, local anesthetic agents of amide type, or any related products (including excipients of the formulations) as well as severe hypersensitivity reactions (like angioedema) to any drugs
* Presence of significant gastrointestinal, liver or kidney disease, or any other conditions known to interfere with the absorption, distribution, metabolism or excretion of drugs or known to potentiate or predispose to undesired effects
* History of significant gastrointestinal, liver or kidney disease that may affect drug bioavailability

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 48 (Actual)
Dates: Start 2022-07-26 (Actual); Primary Completion 2022-08-21 (Actual); Study Completion 2023-05-03 (Estimated)

PRIMARY OUTCOMES:
Cmax between 0 hour to 240 hour after study drug administration | From 0 hour to 240 hour after study drug administration
  Maximum concentration occuring at Tmax
Tmax between 0 hour to 240 hour after study drug administration | From 0 hour to 240 hour after study drug administration
  Time of maximum observed concentration
AUC last | From 0 hour to 240 hour after study drug administration
  Area under the concentration time curve from the time of last dosing to the time of last quantifiable concentration (Tlast)
AUC inf | From 0 hour to 240 hour after study drug administration
  Area under the concentration time curve extrapolated to infinity

CONTACTS AND LOCATIONS:
Overall Officials: Eric Sicard, MD, Principal Investigator — Clinical Research Unit
Locations (1):
- Clinical Research Unit, Montreal, Canada

IPD SHARING:
Plan to Share IPD: No